CLINICAL TRIAL: NCT04597177
Title: Swallowing Sparing IMRT (SW-IMRT) Versus Standard Parotid Sparing IMRT (ST-IMRT) in the Treatment of Head and Neck Cancer
Brief Title: SW-IMRT Versus ST-IMRT in the Treatment of Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD201001409.3
Record Dates: First submitted 2020-09-03; First posted 2020-10-22 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Swallowing Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ST-IMRT (Active Comparator): standard parotid sparing IMRT
  Interventions: Radiation: ST-IMRT SW-IMRT
- SW-IMRT (Experimental): swallowing sparing IMRT
  Interventions: Radiation: ST-IMRT SW-IMRT

INTERVENTIONS:
Radiation: ST-IMRT SW-IMRT

SUMMARY:
To clinically validate whether SW-IMRT actually reduce the occurrence of swallowing dysfunction as compared to ST-IMRT.

DETAILED DESCRIPTION:
Patients are randomly assigned to either ST-IMRT or SW-IMRT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with squamous cell carcinoma and requiring whole neck irradiation as a part of either definitive RT alone or in combination with chemotherapy or post-operative RT either alone or in combination with chemotherapy.

Exclusion Criteria:

* Previous radiotherapy to the head and neck region or prior malignancies, and/or distant metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Subjective assessment of the swallowing function (dysphagia) at regular intervals | 6 months
  Subjective assessment of swallowing function (dysphagia) will be scored on a scale of 0 (no dysphagia) to 4 (life threatening consequences; urgent intervention indicated) each follow-up visit on the basis of National Cancer Institute Common Terminology Criteria for Adverse Events, version 4 (CTCAE 4).
Objective assessment of the swallowing function (dysphagia) at regular intervals | 6 months
  Objective assessment of swallowing will be made by videofluoroscopy and scored by Dynamic Imaging Grade of swallowing toxicity scale (DIGEST) and will be scored on a scale of 0 (no dysphagia) to 4 (life threatening )

SECONDARY OUTCOMES:
local control | 6 months
  Clinical examination and Imaging will be done at regular interval to detect local or nodal recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- May Ashour, Cairo, Egypt